CLINICAL TRIAL: NCT04003584
Title: Is Postoperative Pain Different in the MICS CABG Cohort V. the Traditional Sternotomy Cohort
Brief Title: Postop Pain in the MICS Patients Versus Sternotomy Patients
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB file #09-17-29E
Record Dates: First submitted 2019-06-21; First posted 2019-07-01 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2019-06

CONDITIONS: Pain, Postoperative; Surgery
Keywords: Minimally invasive; Cardiac Surgery; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally Invasive Cardiac Bypass patients
  Interventions: Procedure: Coronary bypass surgery
- Traditional Sternotomy Cardiac Bypass patients
  Interventions: Procedure: Coronary bypass surgery

INTERVENTIONS:
Procedure: Coronary bypass surgery — Reviewed postoperative coronary bypass patients and compared postoperative pain levels

SUMMARY:
To adequately assess postoperative pain in the coronary artery bypass surgical population a multicentered retrospective chart review was carried out; the study utilized a nonexperimental comparative descriptive study design. The retrospective review was conducted over a six-month time frame, consisting of June 2017 through November 2017, at two hospitals within the same organization. The data collection process began in late December of 2017 and January of 2018. The assessment of postop pain was performed by using a standard 11-point numeric pain rating scale on post extubation day one and the day of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an isolated coronary artery bypass surgery at Charlotte Medical Center (CMC) and CMC-Pineville
* Minimally invasive cardiac surgery
* Traditional sternotomy cardiac surgery

Exclusion Criteria:

* Documented history of any chronic pain syndromes requiring active treatment
* The "relative" recent requirement of narcotic analgesic use for pain relief prior to operation
* Any CABG operation that inadvertently resulted in an operative surgical complication
* Patient cases that resulted in a readmission within 30 days from surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective review was conducted over a six-month time frame, consisting of June 2017 through November 2017, at two hospitals within the same organization. One of the hospitals was a level one trauma center in the center of a major southeastern metropolitan area, and the second was a community hospital within the suburbs of the same city's geographic limits. All included patients fit the above inclusion and exclusion criteria per the aforementioned time frame and involved healthcare centers.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Highest reported pain level, on the standard 0-10 pain scale, post extubation day one | The first 24 hours post extubation
  The highest recorded pain level, taken by the nursing staff, on the day following. extubation. Utilized day post due to the washout/possible confounding variable of sedation administration within 24hrs.
Highest reported pain level, on the standard 0-10 pain scale, on the day of discharge. | Within 24 hours from discharge
  The highest reported pain, measured by the nursing staff on within 24hrs from discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jeko Madjarov, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
If requested we would not mind providing guidance on postoperative pain assessments/likert scales.